CLINICAL TRIAL: NCT00615043
Title: A Multi Center Study to Obtain Bladder Tissue Specimens From Subjects Undergoing Transurethral Resection of Bladder Tumor (TURBT) or Other Transurethral Biopsy Procedures
Brief Title: Multi Center Study to Obtain Bladder Tissue Specimens From Patients Undergoing Transurethral Resection Biopsy Procedure
Status: Completed | Type: Observational
Sponsor: Tengion (Industry)
Responsible Party: Sunita Sheth, MD Chief Medical Officer, Tengion, Inc
Other Study IDs: TNG-CL007
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Bladder Disease
Keywords: Transurethral resection of bladder tumor; TURBT
MeSH Terms: conditions — Urinary Bladder Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TURBT group: Subjects undergoing transurethral resection of bladder tumor or other transurethral biopsy procedure who agree to provide bladder tissue specimens
  Interventions: Procedure: Bladder biopsy

INTERVENTIONS:
Procedure: Bladder biopsy — provision of bladder tissue via cystoscopic biopsy during planned TURBT

SUMMARY:
The objective of the study is to obtain bladder tissue specimens from patients otherwise undergoing cystoscopy for use in research at Tengion, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-90 years and undergoing TURBT
* Willing and able to give signed informed consent

Exclusion Criteria:

* Known active infection
* Known colonization with MRSA or VRE
* Receipt of blood or blood products for transfusion during the previous 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients otherwise undergoing TURBT
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of bladder tissue from patients undergoing transurethral resection of bladder tumor or other transurethral biopsy procedure | ongoing throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Sheth, MD, Study Director — Tengion, Inc
Locations (1):
- University of Alabama, Birmingham, Birmingham, Alabama, United States